CLINICAL TRIAL: NCT04305184
Title: A Phase 1/2, Randomized, Placebo-controlled Study to Assess the Safety, Tolerability, Efficacy, and Pharmacokinetics of ASP0598 Otic Solution Following Topical Application Into the Ear in Subjects With Chronic Tympanic Membrane Perforation (CTMP)
Brief Title: A Study to Assess ASP0598 Otic Solution Following Topical Application in the Ear in Subjects With Chronic Tympanic Membrane Perforation (CTMP)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of Efficacy
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 0598-CL-0101
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Results first posted 2024-02-07 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Chronic Tympanic Membrane Perforation
Keywords: ASP0598

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Single Ascending Dose (SAD): 0.03 mcg (Experimental): Participants received single dose of 0.03 microgram (mcg) ASP0598 Otic Solution into the affected ear on day 1 and returned to the investigative site for assessments on days 2, 3, 8, 15, 29, and 57 [End of Study (EOS)].
  Interventions: Drug: ASP0598
- SAD: 0.15 mcg (Experimental): Participants received single dose of 0.15 mcg ASP0598 Otic Solution into the affected ear on Day 1 and returned to the investigative site for assessments on days 2, 3, 8, 15, 29, and 57 (EOS).
  Interventions: Drug: ASP0598
- SAD: 0.75 mcg (Experimental): Participants received single dose of 0.75 mcg ASP0598 Otic Solution into the affected ear on day 1 and returned to the investigative site for assessments on days 2, 3, 8, 15, 29, and 57 (EOS).
  Interventions: Drug: ASP0598
- SAD: 2.25 mcg (Experimental): Participants received single dose of 2.25 mcg ASP0598 Otic Solution into the affected ear on day 1 and returned to the investigative site for assessments on days 2, 3, 8, 15, 29, and 57 (EOS).
  Interventions: Drug: ASP0598
- SAD: Placebo (Placebo Comparator): Participants received single dose of placebo matched to ASP0598 Otic Solution into the affected ear on day 1 and returned to the investigative site for assessments on days 2, 3, 8, 15, 29, and 57 (EOS).
  Interventions: Other: Placebo
- Multiple Ascending Dose (MAD): 0.75 mcg (Experimental): Participants received multiple doses of 0.75 mcg ASP0598 Otic Solution into the affected ear on days 1, 15 and 29 and returned to the investigative site for assessments on days 8, 15, 22, 29, 36, 57, and 85 (EOS).
  Interventions: Drug: ASP0598
- MAD: 2.25 mcg (Experimental): Participants received multiple doses of 2.25 mcg ASP0598 Otic Solution into the affected ear on days 1, 15 and 29 and returned to the investigative site for assessments on days 8, 15, 22, 29, 36, 57, and 85 (EOS).
  Interventions: Drug: ASP0598
- MAD: Placebo (Placebo Comparator): Participants received multiple doses of placebo matched to ASP0598 Otic Solution into the affected ear on days 1, 15 and 29 and returned to the investigative site for assessments on days 8, 15, 22, 29, 36, 57, and 85 (EOS).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ASP0598 — ASP0598 Otic solution was administered onto the Tympanic Membrane (TM) through the external auditory canal via syringe.
  Arms: MAD: 2.25 mcg; Multiple Ascending Dose (MAD): 0.75 mcg; SAD: 0.15 mcg; SAD: 0.75 mcg; SAD: 2.25 mcg; Single Ascending Dose (SAD): 0.03 mcg
Other: Placebo — Placebo matched to ASP0598 Otic solution was administered onto the TM through the external auditory canal via syringe.
  Arms: MAD: Placebo; SAD: Placebo

SUMMARY:
The primary purpose of this study was to evaluate the safety and tolerability of ASP0598 Otic Solution. This study also evaluated the efficacy of ASP0598 otic solution.

DETAILED DESCRIPTION:
This study consisted of a dose escalation (single ascending dose - SAD and multiple ascending dose- MAD) and dose expansion (single dose expansion and/or multiple dose expansion). Dose escalation consisted of up to 4 cohorts for single ascending dose (SAD) and up to 2 cohorts for multiple ascending dose (MAD) with different dose levels. For SAD, after randomization on Day 1, participants received ASP0598 Otic Solution or placebo administration into the affected ear. Participants returned to the site on days 2, 3, 8, 15, 29, and 57 [end of study (EOS)]. Day 3 evaluations were only performed for cohorts 1, 2 and 3. For MAD, after randomization on Day 1, participants received ASP0598 Otic Solution or placebo administration into the affected ear and received additional treatments into the same ear on Days 15 and 29. Participants returned to the investigative site on Days 8, 15, 22, 29, 36, 57, and 85 (EOS). Dose expansion was based on the safety and efficacy results from an interim analysis. An interim analysis was conducted after completion of SAD and again after completion of MAD. The single and multiple dose expansion parts of the study were not opened following review of safety and efficacy results of SAD and MAD parts of the study by the DMC per the Interim Analysis Plan.

ELIGIBILITY:
Inclusion Criteria:

* Subject has chronic tympanic membrane perforation (CTMP) documented as persisting longer than 3 months.
* A female subject is eligible to participate if she is not pregnant and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) OR
  * WOCBP who agrees to follow the contraceptive guidance starting at screening and for at least 28 days after investigational product (IP) application.
* Female subject must agree not to breastfeed starting at drug application on Day 1 and for at least 28 days after IP application.
* Female subject must not donate ova starting on Day 1 and for at least 28 days after investigational product (IP) application.
* A male subject with female partner(s) of child-bearing potential must agree to use contraception starting on Day 1 and for at least 28 days after IP application.
* A male subject must not donate sperm starting on Day 1 and for at least 28 days after IP application.
* Male subject with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom from Day 1 and for at least 28 days after IP application.
* Subject must be willing and able to comply with the study requirements including refraining from using prohibited concomitant medications.
* Subject agrees not to participate in another interventional study during the study period.

Exclusion Criteria:

* Subject has one of following conditions that may affect the ipsilateral side of the ear with chronic tympanic membrane perforation (CTMP):

  * Perforation involving 3 or more quadrants.
  * Pin hole perforation (only for the expansion cohort).
  * Presence of tympanosclerosis adjacent to the perforation.
  * Perforation involves malleus erosion.
  * Absent malleus.
  * Marginal perforation (i.e., involving the annulus or exposing the handle of malleus).
  * Tympanic membrane perforation (TMP) caused by electric/slag/blast/burn injury.
  * Post radiated TMP.
  * History of tympanic membrane repair by any type of live tissue.
  * Active otorrhea or active treatment for otorrhea within the last 3 months prior to Screening.
  * Bellucci otorrhea grade 3 or above.
  * Active external ear canal inflammation (otitis externa, dermatitis) or within the last 3 months prior to Screening.
  * Active diagnosis of Eustachian Tube dysfunction or diagnosis within 6 months prior to Screening.
  * Craniofacial abnormalities, History of head and neck surgery within the last 3 months prior to Screening, history of radiation to head and neck.
  * Recent (within 2 weeks) diagnosis of upper respiratory tract infection.
  * Presence or history of cholesteatoma.
  * Presence of pars-flaccida or pars tensa retraction or adhesion.
  * Presence or history of tumors of the middle or external ear.
  * Contraindications to tympanic membrane closure.
  * An audiometric finding indicates a characteristic of Carhart's notch which is an increase in bone conduction threshold with a peak at 2,000 hertz (Hz).
  * Only hearing ear or better hearing ear and the contralateral ear ≥ 40 dB (decibels) by average four-frequency (500, 1000, 2000 and 4000 Hz).
  * Whole circumference of the tympanic membrane perforation is not visible by endoscope.
  * Presence/history of eosinophilic otitis media in either ear.
* Subject has a presence of adhesive otitis media in the contralateral ear.
* Subject has a presence of any wound healing systemic condition.
* Subject has Obstructive Sleep Apnea where the subject is required to use Continuous Positive Airway Pressure (CPAP) during the study period.
* Subject is exposed in their daily life to high volume of water into the ear canal (e.g., swimmer or surfer).
* Subject has health conditions that would prevent him/her from fulfilling the study requirements on the basis of medical history and laboratory test (Serum Chemistries, complete blood count [CBC] with Differential, Urinalysis) results at the screening visit.
* Subject is receiving any other investigational agents during study participation.
* Subject has any form of substance abuse, or psychiatric illness/social situations that would limit compliance with study requirements, or a condition that could invalidate communication.
* Subject has a known or suspected hypersensitivity to ASP0598, or any components of the formulation used.
* Subject has had previous exposure with ASP0598.
* Subject is unlikely to comply with the visits scheduled in the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (10):
- United States (10):
  - Stanford Hospital, Palo Alto, California
  - Breathe Clear Institute, Torrance, California
  - ENT and Allergy Associates of Florida, Boca Raton, Florida
  - Advanced ENT, New Albany, Indiana
  - Advanced ENT, Louisville, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - Charlotte ENT Associates, Matthews, North Carolina
  - Piedmont ENT, Winston-Salem, North Carolina
  - Carolina ENT Clinic, Orangeburg, South Carolina
  - Richmond ENT, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/0598-CL-0101/
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14533&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with Chronic Tympanic Membrane Perforation (CTMP) documented as persisting longer than 3 months were enrolled in this study.
Pre-assignment Details: Single Ascending Dose (SAD) Multiple Ascending Dose (MAD)
Groups:
- SAD: 0.03 mcg: Participants received single dose of 0.03 microgram (mcg) ASP0598 Otic Solution into the affected ear on day 1 and returned to the investigative site for assessments on days 2, 3, 8, 15, 29, and 57 [End of Study (EOS)].
- MAD: 0.75 mcg: Participants received multiple doses of 0.75 mcg ASP0598 Otic Solution into the affected ear on days 1, 15 and 29 and returned to the investigative site for assessments on days 8, 15, 22, 29, 36, 57, and 85 (EOS).
Period: SAD: Days 1 to 57
Arm/Group | SAD: 0.03 mcg | SAD: 0.15 mcg | SAD: 0.75 mcg | SAD: 2.25 mcg | SAD: Placebo | MAD: 0.75 mcg | MAD: 2.25 mcg | MAD: Placebo
Started | 4 | 4 | 4 | 4 | 4 | 0 | 0 | 0
Completed | 4 | 4 | 4 | 4 | 4 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: MAD: Day 1 to 85
Arm/Group | SAD: 0.03 mcg | SAD: 0.15 mcg | SAD: 0.75 mcg | SAD: 2.25 mcg | SAD: Placebo | MAD: 0.75 mcg | MAD: 2.25 mcg | MAD: Placebo
Started | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF) consisted of all randomized participants who received a dose of study drug.
Groups:
- SAD: 0.03 mcg: Participants received single dose of 0.03 mcg ASP0598 Otic Solution into the affected ear on day 1 and returned to the investigative site for assessments on days 2, 3, 8, 15, 29, and 57 (EOS).
- SAD: ASP0598 0.15 mcg: Participants received single dose of 0.15 mcg ASP0598 Otic Solution into the affected ear on Day 1 and returned to the investigative site for assessments on days 2, 3, 8, 15, 29, and 57 (EOS).
- SAD: ASP0598 0.75 mcg: Participants received single dose of 0.75 mcg ASP0598 Otic Solution into the affected ear on day 1 and returned to the investigative site for assessments on days 2, 3, 8, 15, 29, and 57 (EOS).
- SAD: ASP0598 2.25 mcg: Participants received single dose of 2.25 mcg ASP0598 Otic Solution into the affected ear on day 1 and returned to the investigative site for assessments on days 2, 3, 8, 15, 29, and 57 (EOS).
- MAD: ASP0598 2.25 mcg: Participants received multiple doses of 2.25 mcg ASP0598 Otic Solution into the affected ear on days 1, 15 and 29 and returned to the investigative site for assessments on days 8, 15, 22, 29, 36, 57, and 85 (EOS).
- Total: Total of all reporting groups
Arm/Group | SAD: 0.03 mcg | SAD: ASP0598 0.15 mcg | SAD: ASP0598 0.75 mcg | SAD: ASP0598 2.25 mcg | SAD: Placebo | MAD: 0.75 mcg | MAD: ASP0598 2.25 mcg | MAD: Placebo | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 6 | 6 | 4 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.5 (7.0) | 48.3 (20.4) | 50.8 (7.1) | 49.5 (16.0) | 51.5 (8.1) | 36.5 (18.6) | 44.3 (20.1) | 47.5 (14.0) | 45.11 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 4 | 2 | 2 | 2 | 2 | 1 | 18
  Male | 2 | 1 | 0 | 2 | 2 | 4 | 4 | 3 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 4 | 4 | 3 | 4 | 3 | 6 | 6 | 4 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 4
  White | 4 | 3 | 3 | 3 | 3 | 5 | 5 | 3 | 29
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone Conduction Hearing at 1, 2,4 kilohertz (kHz) by Pure Tone Audiometry (PTA) [Mean (Standard Deviation); unit: decibles] — PTA was a behavioral and quantitative hearing test to assess hearing. Pure tone air conduction and bone conduction tests were used to determine whether there was any unilateral or bilateral hearing loss, what type of hearing loss was present, which frequencies were impacted, and the magnitude of the hearing loss.
  decibles
    1 kHz | 6.3 (7.5) | 6.3 (6.3) | 22.5 (20.2) | 11.3 (11.1) | 12.5 (9.6) | 1.7 (4.1) | 14.2 (15.3) | 3.8 (4.8) | 9.8 (9.9)
    2 kHz | 11.3 (10.3) | 11.3 (7.5) | 25.0 (14.7) | 22.5 (13.2) | 30.0 (21.2) | 10.0 (13.4) | 20.8 (14.6) | 10.0 (5.8) | 17.6 (12.5)
    4 kHz | 6.3 (6.3) | 15.0 (4.1) | 30.0 (24.2) | 28.8 (11.1) | 27.5 (25.3) | 9.2 (17.7) | 21.7 (15.4) | 17.5 (9.6) | 19.5 (14.2)
Tinnitus Visual Analog Scale (TVAS) [Mean (Standard Deviation); unit: Score on a scale] — TVAS was used by participants to rate their tinnitus at baseline and during all subsequent follow-up visits. The scale was a numeric scale and ranged from 0 (not at all strong or loud) to 10 (extremely strong or loud). A lower value indicates less level of discomfort.
  Score on a scale | 1.0 (2.0) | 1.5 (3.0) | 3.0 (3.6) | 3.0 (3.8) | 2.5 (2.9) | 0.7 (1.6) | 3.3 (2.1) | 2.5 (2.1) | 2.2 (2.6)
Ratio of TMP size per total area of tympanic membrane [Mean (Standard Deviation); unit: Percentage of total area of TM] — Ratio of TMP size per total area of tympanic membrane calculation was performed by central imaging vendor and reported as percentage.
  Percentage of total area of TM | 10.3 (5.1) | 11.6 (8.1) | 4.7 (3.8) | 15.8 (11.7) | 7.3 (3.8) | 18.8 (13.4) | 17.1 (9.6) | 8.7 (6.7) | 11.8 (7.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) in SAD
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered an investigational product (IP), and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of IP whether or not considered related to the IP. A TEAE is defined as an AE observed after starting administration of the study drug through end of study visit.
Time Frame: From first dose up to day 57
Population: SAF population
Measure: Number; unit: Participants
Arm/Group | SAD: 0.03 mcg | SAD: 0.15 mcg | SAD: 0.75 mcg | SAD: 2.25 mcg | SAD: Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4
Participants | 4 | 1 | 3 | 3 | 2

2. Primary Outcome: Number of Participants With AE of Special Interest as Cholesteatoma or Ear Neoplasm in SAD
Description: An AE is any untoward medical occurrence in a participant administered an IP, and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of IP whether or not considered related to the IP. Number of participants with cholesteatoma or ear neoplasm is reported.
Time Frame: From first dose up to day 57
Population: SAF population
Measure: Number; unit: Participants
Arm/Group | SAD: 0.03 mcg | SAD: 0.15 mcg | SAD: 0.75 mcg | SAD: 2.25 mcg | SAD: Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4
Participants | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With AE of Special Interest as Ototoxic Symptoms (Tinnitus, Sensorineural Hearing Loss, Dizziness) in SAD
Description: An AE is any untoward medical occurrence in a participant administered an IP, and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of IP whether or not considered related to the IP. Number of participants with any ototoxic symptoms (tinnitus, sensorineural hearing loss, dizziness) is reported.
Time Frame: From first dose up to day 57
Population: SAF population
Measure: Number; unit: Participants
Arm/Group | SAD: 0.03 mcg | SAD: 0.15 mcg | SAD: 0.75 mcg | SAD: 2.25 mcg | SAD: Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4
Participants | 2 | 0 | 1 | 1 | 0

4. Primary Outcome: Number of Participants With AE of Special Interest as Otitis Media or Otitis Externa in SAD
Description: An AE is any untoward medical occurrence in a participant administered an IP, and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of IP whether or not considered related to the IP. Number of participants with otitis media or otitis externa is reported.
Time Frame: From first dose up to day 57
Population: SAF population
Measure: Number; unit: Participants
Arm/Group | SAD: 0.03 mcg | SAD: 0.15 mcg | SAD: 0.75 mcg | SAD: 2.25 mcg | SAD: Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4
Participants | 1 | 0 | 0 | 1 | 0

5. Primary Outcome: Change From Baseline in Bone Conduction Hearing at 1, 2, 4 kHz by Pure Tone Audiometry at Week 8/EOS in SAD
Description: PTA was a behavioral and quantitative hearing test to assess hearing. Pure tone air conduction and bone conduction tests were used to determine whether there was any unilateral or bilateral hearing loss, what type of hearing loss was present, which frequencies were impacted, and the magnitude of the hearing loss.
Time Frame: Baseline and week 8
Population: SAF population
Measure: Mean (Standard Deviation); unit: decibles
Arm/Group | SAD: 0.03 mcg | SAD: 0.15 mcg | SAD: 0.75 mcg | SAD: 2.25 mcg | SAD: Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4
decibles
  1 kHz | -1.3 (2.5) | 0.0 (4.1) | 0.0 (4.1) | -2.5 (6.5) | 1.3 (6.3)
  2 kHz | 1.3 (2.5) | -1.3 (2.5) | 2.5 (8.7) | -3.8 (8.5) | -1.3 (4.8)
  4 kHz | 0.0 (4.1) | -1.3 (4.8) | 1.3 (7.5) | -1.3 (4.8) | 0.0 (7.1)

6. Primary Outcome: Change From Baseline in TVAS at Week 8/EOS in SAD
Description: TVAS was used by participants to rate their tinnitus at baseline and week 8. The scale was a numeric scale and ranged from 0 (not at all strong or loud) to 10 (extremely strong or loud). A lower value indicates less level of discomfort. For the change from baseline, a negative value indicates improvement (less level of discomfort).
Time Frame: Baseline and week 8
Population: SAF population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | SAD: 0.03 mcg | SAD: 0.15 mcg | SAD: 0.75 mcg | SAD: 2.25 mcg | SAD: Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4
Score on a scale | -0.3 (0.5) | 0.0 (0.0) | -1.0 (2.0) | 0.3 (2.9) | -1.5 (2.4)

7. Primary Outcome: Number of Participants With TEAEs in MAD
Description: An AE is any untoward medical occurrence in a participant administered an IP, and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of IP whether or not considered related to the IP. A TEAE is defined as an AE observed after starting administration of the study drug through end of study visit.
Time Frame: From first dose up to day 85
Population: SAF population
Measure: Number; unit: Participants
Arm/Group | MAD: 0.75 mcg | MAD: 2.25 mcg | MAD: Placebo
Number analyzed (Participants) | 6 | 6 | 4
Participants | 6 | 5 | 4

8. Primary Outcome: Number of Participants With AE Special Interest as Cholesteatoma or Ear Neoplasm in MAD
Description: as for outcome 2
Time Frame: From first dose up to day 85
Population: SAF population
Measure: Number; unit: Participants
Arm/Group | MAD: 0.75 mcg | MAD: 2.25 mcg | MAD: Placebo
Number analyzed (Participants) | 6 | 6 | 4
Participants | 0 | 0 | 0

9. Primary Outcome: Number of Participants With AE of Special Interest as Ototoxic Symptoms (Tinnitus, Sensorineural Hearing Loss, Dizziness) in MAD
Description: as for outcome 3
Time Frame: From first dose up to day 85
Population: SAF population
Measure: Number; unit: Participants
Arm/Group | MAD: 0.75 mcg | MAD: 2.25 mcg | MAD: Placebo
Number analyzed (Participants) | 6 | 6 | 4
Participants | 2 | 1 | 0

10. Primary Outcome: Number of Participants With AE of Special Interest as Otitis Media or Otitis Externa in MAD
Description: as for outcome 4
Time Frame: From first dose up to day 85
Population: SAF population
Measure: Number; unit: Participants
Arm/Group | MAD: 0.75 mcg | MAD: 2.25 mcg | MAD: Placebo
Number analyzed (Participants) | 6 | 6 | 4
Participants | 1 | 0 | 0

11. Primary Outcome: Change From Baseline in Bone Conduction Hearing at 1, 2, 4 kHz by Pure Tone Audiometry at Week 12/EOS in MAD
Description: as for outcome 5
Time Frame: Baseline and week 12
Population: SAF population with available data was analyzed.
Measure: Mean (Standard Deviation); unit: decibles
Arm/Group | MAD: 0.75 mcg | MAD: 2.25 mcg | MAD: Placebo
Number analyzed (Participants) | 5 | 6 | 3
decibles
  1 kHz | 1.0 (2.2) | -3.3 (6.1) | -1.7 (2.9)
  2 kHz | 1.0 (2.2) | -2.5 (5.2) | 0.0 (5.0)
  4 kHz | 2.0 (7.6) | -1.7 (6.8) | -6.7 (2.9)

12. Primary Outcome: Change From Baseline in TVAS at Week 12/EOS in MAD
Description: TVAS was used by participants to rate their tinnitus at baseline and week 12. The scale was a numeric scale and ranged from 0 (not at all strong or loud) to 10 (extremely strong or loud). A lower value indicates less level of discomfort. For the change from baseline, a negative value indicates improvement (less level of discomfort).
Time Frame: Baseline and week 12
Population: SAF population with available data was analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MAD: 0.75 mcg | MAD: 2.25 mcg | MAD: Placebo
Number analyzed (Participants) | 5 | 6 | 3
Score on a scale | -0.6 (1.3) | -0.7 (2.0) | 0.0 (2.0)

13. Secondary Outcome: Number of Participants With Complete Closure of Tympanic Membrane Perforation (TMP) at Week 8 for SAD
Description: Tympanic membrane perforation is a hole in the thin membrane that separates the ear canal from the middle ear. TMP closure is defined as microscopic TMP closure without presence of pin hole.
Time Frame: Week 8
Population: The Full Analysis Set (FAS) consisted of all randomized participants who received a dose of study drug and had baseline value and at least 1 post baseline complete closure assessment during study period.
Measure: Number; unit: Participants
Arm/Group | SAD: 0.03 mcg | SAD: 0.15 mcg | SAD: 0.75 mcg | SAD: 2.25 mcg | SAD: Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4
Participants | 0 | 0 | 1 | 0 | 0

14. Secondary Outcome: Number of Participants With Complete Closure of TMP at Week 12 for Dose Expansion
Description: as for outcome 13
Time Frame: Week 12
Population: The single and multiple dose expansion parts of the study were not opened following review of safety and efficacy results of the SAD part of the study by the DMC, therefore the data was not collected.
Arm/Group | SAD: 0.03 mcg | SAD: 0.15 mcg | SAD: 0.75 mcg | SAD: 2.25 mcg | SAD: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Change From Baseline in the Ratio of TMP Size Per Total Area of Tympanic Membrane at Week 8 for SAD
Description: Ratio of TMP size per total area of tympanic membrane calculation was performed by central imaging vendor and measured in percentage.
Time Frame: Baseline and week 8
Population: FAS population with available data was analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of total area of TM
Arm/Group | SAD: 0.03 mcg | SAD: 0.15 mcg | SAD: 0.75 mcg | SAD: 2.25 mcg | SAD: Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 3
Percentage of total area of TM | -0.4 (0.6) | 4.2 (6.3) | -1.8 (2.3) | 1.0 (0.5) | 0.3 (3.0)

16. Secondary Outcome: Change From Baseline in the Ratio of TMP Size Per Total Area of Tympanic Membrane at Week 12 for Dose Expansion
Description: Ratio of TMP size per total area of tympanic membrane calculation was performed by central imaging vendor and was measured by percentage.
Time Frame: Baseline and week 12
Population: as for outcome 14
Arm/Group | SAD: 0.03 mcg | SAD: 0.15 mcg | SAD: 0.75 mcg | SAD: 2.25 mcg | SAD: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Change From Baseline in TMP Size at Week 8 for SAD
Description: TMP size calculation was be performed by central imaging vendor.
Time Frame: Baseline and week 8
Population: FAS population
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | SAD: 0.03 mcg | SAD: 0.15 mcg | SAD: 0.75 mcg | SAD: 2.25 mcg | SAD: Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4
mm^2 | 13451.0 (9700.9) | 14271.5 (11800.6) | 9572.0 (9462.7) | 12784.3 (5277.9) | 27389.0 (37917.3)

18. Secondary Outcome: Change From Baseline in TMP Size at Week 12 for Dose Expansion
Description: TMP size calculation was be performed by central imaging vendor.
Time Frame: Baseline and week 12
Population: as for outcome 14
Arm/Group | SAD: 0.03 mcg | SAD: 0.15 mcg | SAD: 0.75 mcg | SAD: 2.25 mcg | SAD: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Number of Participants With Complete Closure of TMP at Week 12 for MAD
Description: as for outcome 13
Time Frame: Week 12
Population: FAS population
Measure: Number; unit: Participants
Arm/Group | MAD: 0.75 mcg | MAD: 2.25 mcg | MAD: Placebo
Number analyzed (Participants) | 6 | 6 | 4
Participants | 0 | 0 | 1

20. Secondary Outcome: Number of Participants With Complete Closure of TMP at Week 16 for Dose Expansion
Description: as for outcome 13
Time Frame: Week 16
Population: The single and multiple dose expansion parts of the study were not opened following review of safety and efficacy results of the MAD part of the study by the DMC, therefore the data was not collected.
Arm/Group | MAD: 0.75 mcg | MAD: 2.25 mcg | MAD: Placebo
Number analyzed (Participants) | 0 | 0 | 0

21. Secondary Outcome: Change From Baseline in the Ratio of TMP Size Per Total Area of Tympanic Membrane at Week 12 for MAD
Description: as for outcome 15
Time Frame: Baseline and week 12
Population: FAS population
Measure: Mean (Standard Deviation); unit: Percentage of total area of TM
Arm/Group | MAD: 0.75 mcg | MAD: 2.25 mcg | MAD: Placebo
Number analyzed (Participants) | 5 | 6 | 3
Percentage of total area of TM | -0.2 (2.4) | 2.5 (2.3) | 0.3 (2.3)

22. Secondary Outcome: Change From Baseline in the Ratio of TMP Size Per Total Area of Tympanic Membrane at Week 16 for Dose Expansion
Description: as for outcome 15
Time Frame: Baseline and week 16
Population: as for outcome 20
Arm/Group | MAD: 0.75 mcg | MAD: 2.25 mcg | MAD: Placebo
Number analyzed (Participants) | 0 | 0 | 0

23. Secondary Outcome: Change From Baseline in TMP Size at Week 12 for MAD
Description: TMP size calculation was be performed by central imaging vendor.
Time Frame: Baseline and week 12
Population: FAS population with available data was analyzed.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | MAD: 0.75 mcg | MAD: 2.25 mcg | MAD: Placebo
Number analyzed (Participants) | 5 | 6 | 3
mm^2 | 1904.2 (18056.6) | 545.8 (9706.9) | -1237.3 (672.5)

24. Secondary Outcome: Change From Baseline in TMP Size at Week 16 for Dose Expansion
Description: TMP size calculation was be performed by central imaging vendor.
Time Frame: Baseline and week 16
Population: as for outcome 20
Arm/Group | MAD: 0.75 mcg | MAD: 2.25 mcg | MAD: Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: SAD: From first dose up to day 57 MAD: From first dose up to day 85
Description: SAF consisted of all randomized participants who received a dose of study drug in SAD and MAD
Arm/Group | SAD: 0.03 mcg | SAD: ASP0598 0.15 mcg | SAD: ASP0598 0.75 mcg | SAD: ASP0598 2.25 mcg | SAD: Placebo | MAD: 0.75 mcg | MAD: ASP0598 2.25 mcg | MAD: Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/6 | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/6 | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 4/4 | 1/4 | 3/4 | 3/4 | 2/4 | 6/6 | 5/6 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAD: 0.03 mcg (N=4) | SAD: ASP0598 0.15 mcg (N=4) | SAD: ASP0598 0.75 mcg (N=4) | SAD: ASP0598 2.25 mcg (N=4) | SAD: Placebo (N=4) | MAD: 0.75 mcg (N=6) | MAD: ASP0598 2.25 mcg (N=6) | MAD: Placebo (N=4)
Ear canal erythema (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 3 (5) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 5 (11) | 2 (3) | 3 (3)
Ear pruritus (Ear and labyrinth disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Administration site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myringitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Audiogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to limitations of the TM imaging data as evaluated by the central reader, secondary endpoints related to change in TMP size could not be fully evaluated. Following SAD and MAD data review by DMC, the single dose of ASP0598 Otic Solution provided insufficient efficacy to open the single dose expansion study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-08-29): https://cdn.clinicaltrials.gov/large-docs/84/NCT04305184/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT04305184/SAP_001.pdf